CLINICAL TRIAL: NCT06354647
Title: Effectiveness of Zirconia-based Crowns With Retention Grooves (Sprig EZ) Versus Without Retention Grooves (NuSmile ZR) for Restoration of Primary Anterior Teeth: A Parallel-arm Randomized Controlled Trial
Brief Title: Zirconia-based Primary Anterior Crowns With Retention Grooves Versus Without Retention Grooves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20028419
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries; Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconia-based primary anterior crowns with retention grooves (Experimental): Participants will receive zirconia-based primary anterior crowns with retention grooves
  Interventions: Procedure: Zirconia-based primary anterior crowns with retention grooves
- Zirconia-based primary anterior crowns without retention grooves (Experimental): Participants will receive zirconia-based primary anterior crowns without retention grooves
  Interventions: Procedure: Zirconia-based primary anterior crowns without retention grooves

INTERVENTIONS:
Procedure: Zirconia-based primary anterior crowns with retention grooves — Zirconia-based primary anterior crowns with retention grooves
  Arms: Zirconia-based primary anterior crowns with retention grooves
Procedure: Zirconia-based primary anterior crowns without retention grooves — Zirconia-based primary anterior crowns without retention grooves
  Arms: Zirconia-based primary anterior crowns without retention grooves

SUMMARY:
The purpose of this research study is to test the effectiveness of two different crowns/caps on teeth for restoration of primary anterior teeth. The two different materials of crowns are esthetic crowns with retentive grooves and without retentive crowns. These crowns are placed on the teeth to restore function, esthetics and prevent further caries and infection.

DETAILED DESCRIPTION:
There are many treatment options available for restoring primary anterior teeth. A clinician's decision to opt for any specific treatment option is based on multiple factors such as the clinician's liking of a specific material or method, esthetic demands by parents, the child's behavior, and moisture and hemorrhage control. Out of many treatment options, preformed zirconia crowns for primary teeth have been available for over a decade. There is insufficient research that compares the success of anterior pediatric zirconia crowns with and without retentive grooves.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 2 to 6-year-old children.
* Those having opposed anterior teeth.
* No history of systemic illness or dental developmental anomalies
* Minimal of two surfaces of caries in the upper anterior teeth.
* Patient with Early Childhood Caries.
* Patients treated under General Anesthesia.
* English, Spanish, and Arabic speaking patients

Exclusion Criteria:

* Teeth nearing exfoliation.
* The presence of a single surface caries, not involving the proximal surfaces.
* Teeth that have been subjected to trauma.
* Bruxism.
* Special health needs.
* Presence of teeth wear on the opposing teeth, or absence of opposing teeth.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Success of prefabricated Zirconia-based primary anterior crowns with retention grooves compared to Zirconia-based primary anterior crowns without retention grooves through clinical outcomes | 3, 6, 12, 24 and 36 months
  The clinical outcomes will be measured and reported in the data table based on the number of participants scored on 3-point Likert scale (Ideal, Acceptable, or Not Acceptable) for the following parameters separately:
  Contour of crown, Gingival health, Staining of crown, Surface roughness of crown, Opposing tooth, Color match of crown, Marginal fit, Marginal discoloration, Recurrent caries.
Success of prefabricated Zirconia-based primary anterior crowns with retention grooves compared to Zirconia-based primary anterior crowns without retention grooves through radiographic outcomes | 3, 6, 12, 24 and 36 months
  The radiographic outcomes will be measured and reported in the data table based on the number of participants scored on either presence or absence (yes/no) of the findings for the following parameter separately: Widening of periodontal ligament space, periapical pathology, alveolar crestal bone loss, internal root resorption and external root resorption.

SECONDARY OUTCOMES:
Parental satisfaction | 3, 12, 24 and 36 months
  The questionnaire is a Likert scale of 1-5. 1 equals very dissatisfied. 5 equals very satisfied. The higher the score, the better.
Child satisfaction | 3, 12, 24 and 36 months
  The questionnaire is a Likert scale of 1-5. 1 equals very dissatisfied. 5 equals very satisfied. The higher the score, the better.
Oral health impact during early childhood | 3, 12, 24 and 36 months
  Evaluating Oral health impact during early childhood utilizing the Early Childhood Oral Health Impact Scale (ECOHIS) questionnaire. This is rated on a Likert 5-point scale. (0 = never, 1 = hardly ever, 2 = occasionally, 3 = often, 4 = very often)

CONTACTS AND LOCATIONS:
Overall Officials: Jayakumar Jayaraman, MDS, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No